CLINICAL TRIAL: NCT01738373
Title: Investigator Centers Will Be All French Hematology Centers Performing Autologous Transplantation and Prescribing Mozobil in Hematopoietic Stem Cell Mobilization Willing to Participate In This Study
Brief Title: Registry of Patients Treated With Plerixafor (Mozobil®) for Haematopoietic Stem Cell Mobilization Before Autologous Transplantation
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MOZ22510
Record Dates: First submitted 2012-11-26; First posted 2012-11-30 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Bone Marrow / Autologous Transplants
Keywords: autologous stem cell transplantation; lymphoma; multiple myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — plerixafor

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Plerixafor — Plerixafor will be prescribed independently by the physician, according to usual practice.
  Other Names: Mozobil®

SUMMARY:
The aim of this registry is to provide information, in day-to-day practice, on Plerixafor prescription modalities in France, over a 13-month period in order to address the health authorities' request.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Plerixafor for autologous transplantation between November 2011 and November 2012
* Patients who have been informed and who have given their written consent for the access to their medical file

Exclusion Criteria:

* Patients already included in a Plerixafor ongoing clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The selection of the registry's participants will be based on an exhaustive request of all apheresis centers distributed in the French territory.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The characteristics of the patients who received treatment | 13 months
Dosage of treatment | 13 months
Number of CD34+ cells collected following treatment | 13 months
Number of patients with the existence of one or more predictive factors of poor mobilisation | 13 months
Duration of treatment | 13 months
Associated treatments | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Marseille, France